CLINICAL TRIAL: NCT01064622
Title: A Multi-center, Double Blind, Placebo-Controlled, Randomized Phase II Trial of Gemcitabine Plus GDC-0449 (NSC 747691), a Hh Pathway Inhibitor, in Patients With Metastatic Pancreatic Cancer (10052747)
Brief Title: Gemcitabine Hydrochloride With or Without Vismodegib in Treating Patients With Recurrent or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2011-01454; NCI-2011-01454 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10-00099; CDR0000655378; UCCRC-8418; 09-068 (Other: University of Chicago Comprehensive Cancer Center); 8418 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); N01CM62201 (NIH); N01CM62204 (NIH); N01CM62209 (NIH); P30CA014599 (NIH)
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Results first posted 2015-02-13 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Adenocarcinoma; Recurrent Pancreatic Carcinoma; Stage IV Pancreatic Cancer AJCC v6 and v7
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Hydrocortisone; HhAntag691

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (gemcitabine hydrochloride and placebo) (Active Comparator): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and placebo PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. At the time of disease progression, patients are unblinded and may crossover to arm II.
  Interventions: Drug: Gemcitabine Hydrochloride; Other: Hydrocortisone/Placebo
- Arm II (gemcitabine hydrochloride and vismodegib) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and vismodegib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Gemcitabine Hydrochloride; Drug: Vismodegib

INTERVENTIONS:
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011
Other: Hydrocortisone/Placebo — Given PO
  Other Names: Hydrocortisone Used as a Placebo
  Arms: Arm I (gemcitabine hydrochloride and placebo)
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC 0449; GDC-0449; GDC0449; Hedgehog Antagonist GDC-0449
  Arms: Arm II (gemcitabine hydrochloride and vismodegib)

SUMMARY:
This randomized phase I/II trial studies gemcitabine hydrochloride and vismodegib to see how well they work compared with gemcitabine hydrochloride alone in treating patients with recurrent or metastatic pancreatic cancer. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vismodegib may slow the growth of tumor cells. It is not yet known whether giving gemcitabine hydrochloride together with vismodegib is more effective than gemcitabine hydrochloride alone in treating patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To compare the progression-free survival of advanced pancreatic cancer patients treated with the combination of gemcitabine plus GDC-0449 (vismodegib) versus gemcitabine plus placebo.

SECONDARY OBJECTIVES:

I. To compare overall survival of advanced pancreatic cancer patients treated with the combination of gemcitabine plus GDC-0449 versus gemcitabine plus placebo.

II. To compare the objective response rate of advanced pancreatic cancer patients treated with the combination of gemcitabine plus GDC-0449 versus gemcitabine alone.

III. To determine the toxicity experienced by pancreatic cancer patients treated with the combination of gemcitabine plus GDC-0449.

IV. To determine the activity, in an exploratory analysis, of gemcitabine plus GDC-0449 in patients who progress on gemcitabine plus placebo.

TERTIARY OBJECTIVES:

I. To determine if tumor immunohistochemical expression patterns of proteins in the Hh pathway, including sonic hedgehog (Shh), indian hedgehog (Ihh), patched tumor suppressor gene (PTCH), smoothened protein (SMO), and GLI1 and 2, within pancreatic tissue obtained at the time of curative intent surgery predict response and prognosticate outcome of patients treated with or without GDC-0449 at the time of relapse.

II. To determine the prognostic ability (relapse free survival, [RFS]) of these biologic markers for resected patients in an archival cohort of patients undergoing resection.

III. To determine expression pattern of pancreatic CSC markers, including CD44, CD24, CD133, aldehyde dehydrogenase (ALDH) and epithelial specific antigen (ESA) by immunohistochemistry (IHC) on these archival tissues in relation to Hh pathway markers and correlate these with clinical outcomes.

IV. To determine whether high baseline serum Shh, as well as changes in serum Shh during treatment, predict treatment efficacy and/or prognosticate clinical outcome.

V. To determine the frequency of mutation of Hh pathway genes, PTCH, SMO, SuFU, and if the presence or absence of mutations are correlated with clinical outcome.

VI. To determine the frequency of amplification of Hh pathway genes, gene copy number by quantitative polymerase chain reaction (qPCR) of GLI1 and SMO in those tumors that have high protein expression as seen by IHC. Gene amplification will be correlated with clinical outcome.

VII. To determine if there is a correlation of K-ras mutation, and MET and RON expression, amplification, or mutation status with Hh pathway abnormalities, CSC markers, and clinical outcomes.

VIII. To determine if baseline contrast perfusion imaging volume transfer constant (Ktrans) within primary and liver metastatic lesions as measured on a 256-detector computed tomography (CT) scanner predicts objective response rates, and other clinical endpoints including progression-free survival (PFS), to treatment with gemcitabine and GDC-0449/placebo. (University of Chicago ONLY) IX. To determine if treatment with Gemcitabine and GDC-0449 improves tumor perfusion, as measured by Ktrans, over the course of treatment by serial CT scans every 2 cycles, compared to tumors treated with Gemcitabine and placebo. (University of Chicago ONLY) X. To determine if improved tumor perfusion with GDC-0449 treatment (if observed) improves objective response rates and other clinical endpoints including PFS. (University of Chicago ONLY)

OUTLINE: This is a multicenter, safety lead-in study (part I) followed by a randomized study (part II).

An initial 6 patients are enrolled in the part I portion of the study. If no dose-limiting toxicities occur in these patients, subsequent patients are enrolled in the part II portion of the study.

PART I (safety lead-in study): Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15 and hedgehog antagonist GDC-0449 orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PART II (randomized study): Patients are stratified according to disease status (recurrent after surgery vs metastatic) and Eastern Cooperative Oncology Group (ECOG) performance status (0 vs 1). Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive gemcitabine hydrochloride 1000 mg/m^2 IV over 30 minutes on days 1, 8, and 15 and placebo PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. At the time of disease progression, patients are unblinded and may crossover to arm II.

ARM II: Patients receive gemcitabine hydrochloride 1000 mg/m^2 IV over 30 minutes on days 1, 8, and 15 and hedgehog antagonist GDC-0449 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Tumor tissue, blood, serum, and plasma samples are collected periodically for biomarker and other analyses.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the pancreas
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients must have either:

  * Newly diagnosed chemo-naïve metastatic pancreatic cancer; only patients who have not received any chemotherapy for their metastatic disease are eligible
  * Recurrent disease after curative-intent surgery which has now recurred and is metastatic; patients who have recurrent disease may have received adjuvant chemotherapy or adjuvant chemoradiation, but may not have received any chemotherapy for metastatic disease; adjuvant therapy must have been completed >= 6 months prior to the diagnosis of recurrent disease, or if not adjuvant therapy received, surgery must have been performed >= 6 months prior to the diagnosis of recurrent disease
* Age >= 21 years
* Life expectancy > 3 months
* Karnofsky performance status >= 80%
* Granulocytes >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Total bilirubin =< 1.5 times upper limit of normal (ULN)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 times upper limit of normal (ULN) (=< 5 times ULN in the presence of liver metastases)
* Creatinine within normal institutional limit (< 1.5) OR creatinine clearance >= 65 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* International normalized ratio (INR) =< 1.5 (=< 3 for patients on warfarin)
* Patients who are on warfarin anticoagulation are allowed to participate as long as they fit the following 4 criteria:

  * They are therapeutic on a stable warfarin dose
  * Their INR target range is no greater than 3
  * They are monitored with weekly INR testing
  * They have no active bleeding or pathological condition that carries high risk of bleeding Other anticoagulants, including enoxaparin (Lovenox) and fondaparinux (Arixtra) are also permitted
* Women of child-bearing potential and men must use at least one form of contraception (i.e., barrier contraception) at least 4 weeks prior to study entry and then two forms of contraception (i.e barrier contraception and one other method of contraception), for the duration of study participation, and for at least 12 months post-treatment; for appropriate methods of contraception considered acceptable; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Pregnancy Testing: Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days (at initial screening/consideration for the trial - serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of GDC-0449; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing GDC-0449, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of GDC-0449
* Ability to understand and the willingness to sign a written informed consent document
* Patients with recurrent disease after curative-intent surgical resection must have sufficient archival material for correlative studies (20 unstained 5 micron slides and 20 unstained 10 micron slides, or an archival tissue block

Exclusion Criteria:

* No prior chemotherapy for metastatic pancreatic cancer; patients who have received any chemotherapy and/or radiation therapy in the adjuvant setting must have completed this therapy ≥6 months prior to enrollment on the trial at the time of recurrence
* Patients may not be receiving (or received prior to enrollment) any other investigational agents for metastatic disease
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to hedgehog antagonist GDC-0449 or any other agents used in this study
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or other agents used in the study
* GDC-0449 inhibits CYP2C8, CYP2C9, and CYP2C19 drug metabolism enzymes in vitro at concentrations that may be clinically relevant. Therefore, caution should be exercised when dosing GDC-0449 concurrently with medications that are substrates of CYP2C8, CYP2C9, and CYP2C19 and have narrow therapeutic windows
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow capsules
* Patients with clinically active liver disease, including active viral or other hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia, defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* No currently active second malignancy other than non-melanoma skin cancer or carcinoma in-situ of the cervix; patients are not considered to have a "currently active" malignancy if they have completed therapy and have no evidence of recurrence for at least 5 years
* Uncontrolled intercurrent illness including, but not limited to,

  * Ongoing or active infection,
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GDC-0449; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with GDC-0449; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-09-03 (Actual); Primary Completion 2012-12-09 (Actual); Study Completion 2013-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L Kindler, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (25):
- United States (25):
  - Tower Cancer Research Foundation, Beverly Hills, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Catenacci DV, Junttila MR, Karrison T, Bahary N, Horiba MN, Nattam SR, Marsh R, Wallace J, Kozloff M, Rajdev L, Cohen D, Wade J, Sleckman B, Lenz HJ, Stiff P, Kumar P, Xu P, Henderson L, Takebe N, Salgia R, Wang X, Stadler WM, de Sauvage FJ, Kindler HL. Randomized Phase Ib/II Study of Gemcitabine Plus Placebo or Vismodegib, a Hedgehog Pathway Inhibitor, in Patients With Metastatic Pancreatic Cancer. J Clin Oncol. 2015 Dec 20;33(36):4284-92. doi: 10.1200/JCO.2015.62.8719. Epub 2015 Nov 2. PMID 26527777

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to the phase II randomized trial, an open-label, lead-in phase I study was conducted with all patients receiving gemcitabine hydrochloride plus vismodegib. Seven patients were enrolled and no safety issues were identified.
Period: Lead-in Phase I
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib)
Started | 0 | 7
Completed | 0 | 7
Not Completed | 0 | 0
Period: Randomized Phase II
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib)
Started | 55 | 56
Completed | 53 | 53
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 0 | 1
Period: Crossover of Arm I
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib)
Started | 22 (Among 53 patients, 45 had disease progression; however 23 elected not to crossover to vismodegib.) | 0
Completed | 22 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I lead-in Patients: Patients enrolled in the lead-in phase I portion of the trial. Patients receive 1000 mg/m2 gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and 150 mg vismodegib PO QD on days 1-28.
- Total: Total of all reporting groups
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients | Total
Number analyzed (Participants) | 53 | 53 | 7 | 113
Age, Continuous [Mean (Full Range); unit: years] — One age value missing from Arm I.
  years | 64.5 [39 to 84] | 64.7 [49 to 82] | 56.7 [43 to 72] | 64.1 [39 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 2 | 50
  Male | 27 | 31 | 5 | 63
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 0 | 16
  White | 45 | 40 | 7 | 92
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Time from randomization to disease progression or death from any cause. Estimated in the two treatment groups by the Kaplan-Meier method and compared using a stratified logrank test.
Time Frame: Up to 3 years
Population: Phase I lead-in patients were not included in the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase I lead-in Patients: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and vismodegib PO QD on days 1-28.
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients
Number analyzed (Participants) | 53 | 53 | 0
months | 2.5 [1.9 to 3.8] | 4.0 [2.5 to 5.3] |
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride and Placebo) vs Arm II (Gemcitabine Hydrochloride and Vismodegib); Test type: Superiority or Other; p = 0.15, Log Rank — Reported p-value is one-sided. p<0.10 required for statistical significance; Stratified by Karnofsky performance status (90-100 vs. 80) and disease status (newly diagnosed vs. recurrent after surgery); Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.55 to 1.22] — Hazard ratio is for (gemcitabine hydrochloride plus vismodegib)/(gemcitabine hydrochloride plus placebo), adjusted for Karnofsky performance status (90-100 vs. 80) and disease status (newly diagnosed vs. recurrent after surgery)

2. Secondary Outcome: Overall Survival
Description: Time from randomization to death from any cause. Estimated in the two treatment groups by the Kaplan-Meier method and compared using a stratified logrank test.
Time Frame: Up to 3 years
Population: Phase I lead-in patients were not included in the efficacy analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients
Number analyzed (Participants) | 53 | 53 | 0
months | 6.1 [5.0 to 8.1] | 6.9 [5.8 to 8.0] |
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride and Placebo) vs Arm II (Gemcitabine Hydrochloride and Vismodegib); Test type: Superiority or Other; p = 0.37, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.64 to 1.46] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months
Population: Phase I lead-in patients were not included in the efficacy analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients
Number analyzed (Participants) | 53 | 53 | 0
percentage of participants | 13.2 [5.5 to 25.3] | 7.5 [2.1 to 18.2] |
Statistical Analysis 1: Comparison: Arm I (Gemcitabine Hydrochloride and Placebo) vs Arm II (Gemcitabine Hydrochloride and Vismodegib); Test type: Superiority or Other; p = 0.42, Cochran-Mantel-Haenszel — Two-sided p-value for Cochran-Mantel-Haenszel test stratified by Karnofsky performance status and disease status

4. Secondary Outcome: Incidence of Adverse Events
Description: Details are provided in Adverse Events section below. Reported here are percentage of patients in each arm with any grade 1 or higher adverse event, regardless of attribution.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients
Number analyzed (Participants) | 53 | 53 | 7
percentage of participants | 98.1 [89.9 to 99.9] | 98.1 [89.9 to 99.9] | 100.0 [59.0 to 100.0]

5. Secondary Outcome: Activity (Overall Response Rate) in Crossover Patients
Description: RECIST response rate in patients after crossover from placebo to vismodegib arm. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months
Population: Phase I lead-in patients were not included in the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients
Number analyzed (Participants) | 22 | 0 | 0
percentage of participants | 4.5 [0.1 to 22.8] |  |

ADVERSE EVENTS:
Time Frame: Up to 3 years.
Groups:
- Phase II Crossover Patients: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and vismodegib PO QD on days 1-28.
Arm/Group | Arm I (Gemcitabine Hydrochloride and Placebo) | Arm II (Gemcitabine Hydrochloride and Vismodegib) | Phase I lead-in Patients | Phase II Crossover Patients
Serious Adverse Events (participants affected / at risk) | 37/53 | 22/53 | 5/7 | 4/22
Other Adverse Events (participants affected / at risk) | 52/53 | 52/53 | 7/7 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gemcitabine Hydrochloride and Placebo) (N=53) | Arm II (Gemcitabine Hydrochloride and Vismodegib) (N=53) | Phase I lead-in Patients (N=7) | Phase II Crossover Patients (N=22)
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Death due to disease progression (General disorders) | 1 | 0 | 0 | 0
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L): Urinary tract NOS (Infections and infestations) | 1 | 0 | 0 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils: Blood (Infections and infestations) | 0 | 1 | 0 | 0
Metastatic Pancreatic Cancer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
cholestasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
disease progression (Gastrointestinal disorders) | 1 | 0 | 0 | 0
failure to thrive (General disorders) | 0 | 1 | 0 | 1
neoplasmsbenign, malignant and unspecified (Gastrointestinal disorders) | 1 | 0 | 0 | 0
progression of disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0
progression of metastatic pancreatic cancer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
progressive disease (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 6 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 0
Creatinine increased (Investigations) | 1 | 1 | 0 | 0
Death NOS (General disorders) | 6 | 4 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Fever (General disorders) | 4 | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Hallucinations (Psychiatric disorders) | 1 | 0 | 0 | 0
Hepatic infection (Infections and infestations) | 0 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
INR increased (Investigations) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1 | 0 | 0
Jejunal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 2 | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 4 | 0 | 0
Nervous system disorders - Other (Nervous system disorders) | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 3 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Peripheral ischemia (Vascular disorders) | 0 | 1 | 0 | 0
Peritoneal infection (Infections and infestations) | 2 | 0 | 0 | 0
Platelet count decreased (Investigations) | 2 | 3 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 4 | 2 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3 | 2 | 0
Weight loss (Investigations) | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 — NOS
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Gemcitabine Hydrochloride and Placebo) (N=53) | Arm II (Gemcitabine Hydrochloride and Vismodegib) (N=53) | Phase I lead-in Patients (N=7) | Phase II Crossover Patients (N=22)
Abdominal pain (Gastrointestinal disorders) | 19 | 10 | 3 | 6
Agitation (Psychiatric disorders) | 0 | 3 | 0 | 0
Alanine aminotransferase increased (Investigations) | 27 | 28 | 6 | 9
Alkaline phosphatase increased (Investigations) | 23 | 25 | 6 | 11
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 8 | 2 | 0
Anemia (Blood and lymphatic system disorders) | 41 | 40 | 6 | 17
Anorexia (Metabolism and nutrition disorders) | 18 | 20 | 5 | 9
Anxiety (Psychiatric disorders) | 3 | 3 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 4 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 29 | 25 | 4 | 13
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 1 | 3
Blood bilirubin increased (Investigations) | 12 | 11 | 2 | 6
Chills (General disorders) | 8 | 6 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 3 | 0 | 0
Constipation (Gastrointestinal disorders) | 14 | 17 | 5 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 1 | 0
Creatinine increased (Investigations) | 6 | 5 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 10 | 6 | 0 | 2
Depression (Psychiatric disorders) | 1 | 5 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 12 | 13 | 0 | 3
Dizziness (Nervous system disorders) | 4 | 6 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 12 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 5 | 4 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 0 | 3
Edema limbs (General disorders) | 13 | 9 | 1 | 0
Fatigue (General disorders) | 36 | 37 | 5 | 12
Fever (General disorders) | 7 | 12 | 1 | 4
Flatulence (Gastrointestinal disorders) | 5 | 5 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 | 6 | 0 | 0
General disorders and administration site conditions - Other (General disorders) | 5 | 7 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 0
Headache (Nervous system disorders) | 7 | 10 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 26 | 28 | 4 | 11
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 7 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 3 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 30 | 24 | 2 | 14
Hypocalcemia (Metabolism and nutrition disorders) | 21 | 17 | 3 | 7
Hypoglycemia (Metabolism and nutrition disorders) | 3 | 5 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 12 | 17 | 2 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 12 | 13 | 2 | 2
Hyponatremia (Metabolism and nutrition disorders) | 21 | 16 | 4 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 6 | 7 | 0 | 0
Hypotension (Vascular disorders) | 3 | 4 | 0 | 2
Infections and infestations - Other (Infections and infestations) | 0 | 4 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 5 | 1 | 0
Investigations - Other (Investigations) | 3 | 5 | 0 | 0
Lymphocyte count decreased (Investigations) | 17 | 9 | 0 | 7
Mucositis oral (Gastrointestinal disorders) | 3 | 3 | 0 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 2
Nausea (Gastrointestinal disorders) | 29 | 29 | 5 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 0 | 0
Neutrophil count decreased (Investigations) | 25 | 28 | 3 | 6
Pain (General disorders) | 6 | 14 | 2 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 10 | 1 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 7 | 0 | 3
Platelet count decreased (Investigations) | 30 | 32 | 6 | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 5 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 6 | 4 | 0 | 2
Syncope (Nervous system disorders) | 3 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 4 | 3 | 1 | 0
Vascular disorders - Other (Vascular disorders) | 1 | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 18 | 19 | 5 | 5
Weight loss (Investigations) | 10 | 11 | 0 | 0
White blood cell decreased (Investigations) | 31 | 27 | 5 | 9
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 1 | 0
Cancer pain (General disorders) | 0 | 0 | 1 | 0
Death NOS (General disorders) | 0 | 0 | 7 | 0
Dysphagia, esophagiti9s, odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Renal and urinary disorders, other (Renal and urinary disorders) | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less